CLINICAL TRIAL: NCT02946255
Title: Testing the Effectiveness of a Brief, Peer Support Intervention to Facilitate Transition Form Psychiatric Hospitalization
Brief Title: Testing the Effectiveness of The Welcome Basket Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Sean Kidd, Independent Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 073/2016
Record Dates: First submitted 2016-10-12; First posted 2016-10-27 (Estimated); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-08

CONDITIONS: Psychosis
Keywords: Psychosis; Psychosis NOS; Schizophrenia; Hospital discharge; Inpatient psychiatry
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders; Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Welcome Basket Brief (WBbr) (Experimental): The brief version of the Welcome Basket (WBbr) was developed based upon the observation in feasibility testing that for some participants much of the benefit of this approach appeared to be centred upon the visits immediately prior and subsequent to discharge. In the WBbr the same core components will be present, albeit in an abbreviated form with one 30-60 minute visit in the week prior to discharge and a single, 3-hour visit in the week subsequent to discharge in which the welcome basket would be delivered, core CAT strategies discussed and implemented, and some basic orientation to community resources undertaken. This brief version of the intervention has not to date been studied.
  Interventions: Behavioral: Welcome Basket Brief (WBbr)
- Welcome Basket (WB) (Experimental): Peer Support Workers (PSWs) hold 1-2 meetings with clients (30-60 minutes) in the 2-week period before they are discharged from hospital. They describe the program and undertake an assessment. From this assessment the two core components of the intervention are initiated. First, a "welcome basket" is created for the client. The PSW also forms a plan with the client about tours of their neighbourhood to familiarize them with the local resources and support them in building confidence in accessing their local communities. These activities will take place through weekly visits (2 hours/visit) in the 4 weeks immediately following discharge. WB will be provided in combination with core Cognitive Adaptation Training (CAT) compensatory interventions.
  Interventions: Behavioral: Welcome Basket (WB)
- Treatment As Usual (Active Comparator): Treatment as usual (TAU) involves the typical discharge procedures for clients from Unit 2, Forensic and EPU wards at CAMH. It includes referral to outpatient psychiatric services and relevant community supports with the transition facilitated by inpatient social work staff.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Welcome Basket (WB) — Peer Support Workers (PSWs) hold 1-2 meetings with clients (30-60 minutes) in the 2-week period before they are discharged from hospital. They describe the program and undertake an assessment. From this assessment the two core components of the intervention are initiated. First, a "welcome basket" is created for the client. The PSW also forms a plan with the client about tours of their neighbourhood to familiarize them with the local resources and support them in building confidence in accessing their local communities. These activities will take place through weekly visits (2 hours/visit) in the 4 weeks immediately following discharge. WB will be provided in combination with core Cognitive Adaptation Training (CAT) compensatory interventions.
  Arms: Welcome Basket (WB)
Behavioral: Welcome Basket Brief (WBbr) — The brief version of the Welcome Basket (WBbr) was developed based upon the observation in feasibility testing that for some participants much of the benefit of this approach appeared to be centred upon the visits immediately prior and subsequent to discharge. In the WBbr the same core components will be present, albeit in an abbreviated form with one 30-60 minute visit in the week prior to discharge and a single, 3-hour visit in the week subsequent to discharge in which the welcome basket would be delivered, core CAT strategies discussed and implemented, and some basic orientation to community resources undertaken. This brief version of the intervention has not to date been studied.
  Arms: Welcome Basket Brief (WBbr)
Behavioral: Treatment As Usual — Treatment as usual (TAU) involves the typical discharge procedures for clients from Unit 2, Forensic and EPU wards at CAMH. It includes referral to outpatient psychiatric services and relevant community supports with the transition facilitated by inpatient social work staff.
  Arms: Treatment As Usual

SUMMARY:
The investigators propose to examine the effectiveness of a brief intervention that might better facilitate the transition into the community for people with schizophrenia or bipolar disorder with psychotic features. The intervention is called the Welcome Basket. It involves Peer Support Workers connecting with and supporting hospitalized individuals in the days before discharge and again in the community in the first month immediately following discharge. The investigators will compare the outcomes of discharge from hospital as usual with the full version of the welcome basket and a preliminary test of an abbreviated 2 visit version of the intervention.

DETAILED DESCRIPTION:
Discharge from hospital has been highlighted as a critical time in the care of individuals with mental illness. The peak period of risk for readmission for individuals with severe mental illness is in the first month and the highest risk for post-discharge suicide is within the first 2 weeks with discontinuity of contact with providers highlighted as a key risk factor. One half of individuals with schizophrenia miss their first-scheduled outpatient appointment following discharge and this time is a key period of risk for medication non-compliance. Common problems that occur at the time of discharge from psychiatric care settings include poor communication between inpatient and outpatient providers and inadequate involvement and support of families. The research literature on effective practices linked with discharge is strikingly sparse given the evidence that this is a period of heightened risk.

The investigators hypothesize that the Welcome Basket intervention will improve the discharge-related outcomes of individuals with schizophrenia or bipolar disorder with psychotic features compared to treatment as usual. Investigators will also explore the outcomes of an abbreviated, 2-visit version of the intervention. This study will employ a randomized, controlled trial design. Inpatient clients with a diagnosis of schizophrenia spectrum mental illness or bipolar disorder with psychotic features will be randomized with a 2:2:1 ratio to: treatment as usual, the full welcome basket intervention, and the abbreviated intervention. Measures will include re-hospitalization, symptomatology, quality of life, and community functioning. Assessments at baseline, 4 weeks post-discharge, and 6 months post-discharge will facilitate studies of relative effectiveness and sustainment of gains. This design will facilitate an examination of both overall outcomes as well as some preliminary dismantling of mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be adults, 18 years of age or older, with a chart diagnosis of a schizophrenia spectrum mental illness or bipolar disorder with psychotic features confirmed by Module B (psychotic symptoms) of the Structured Clinical Interview for DSM-5 (SCID-5) (First, William, Karg, & Spitzer, 2015). All participants will be on CAMH inpatient units at the time of recruitment and will have been in continuous inpatient care for close to or more than 2 weeks. This timeframe is guided by the rationale and experience indicating that an overly brief period of hospitalization circumscribes the relevance of the intervention.
2. Participants will be returning to places of residence in the Greater Toronto Area (catchment of CAMH) or can travel to the GTA if they will reside outside the catchment area.
3. Participants must have been referred to outpatient case management.
4. Proposed housing arrangements must be stable and conducive to the intervention. If homelessness or emergency shelter residence appears likely, or boarding home policy precludes any external staff from entering the premises, such individuals will be excluded.
5. Proficiency in English.

Exclusion criteria:

1. Do not meet the above criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean A Kidd, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barker S, Barron N, McFarland BH, Bigelow DA. A community ability scale for chronically mentally ill consumers: Part I. Reliability and validity. Community Ment Health J. 1994 Aug;30(4):363-83. doi: 10.1007/BF02207489. PMID 7956112
- [Background] Lee, K., Brekke, J., Yamada, A., & Chou, C. (2010). Longitudinal invariance of the satisfaction with life scale for individuals with schizophrenia. Research on Social Work Practice, 20(2), 234-241.
- [Background] Derogatis, L.R.(1993). BSI Brief Symptom Inventory: Administration, Scoring, and Procedure Manual (4th Ed.). Minneapolis, MN: National Computer Systems.
- [Background] Barbic, S., Kidd, SA, Backman, C., MacEwan, W.. Honer, W., & McKenzie, K. (2016). The development and testing of the Personal Recovery Outcome Measure (PROM) [in preparation].
- [Background] Stergiopoulos V, Gozdzik A, Misir V, Skosireva A, Connelly J, Sarang A, Whisler A, Hwang SW, O'Campo P, McKenzie K. Effectiveness of Housing First with Intensive Case Management in an Ethnically Diverse Sample of Homeless Adults with Mental Illness: A Randomized Controlled Trial. PLoS One. 2015 Jul 15;10(7):e0130281. doi: 10.1371/journal.pone.0130281. eCollection 2015. PMID 26176621
- [Background] First MB, William JBW, Karg RS, Spitzer RL: Structured Clinical Interview for DSM-5-Research Version (SCID-5 for DSM-5, Research Version; SCRID-5-RV). Arlington,VA, American Psychiatric-Association, 2015.
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Dennis ML, Chan YF, Funk RR. Development and validation of the GAIN Short Screener (GSS) for internalizing, externalizing and substance use disorders and crime/violence problems among adolescents and adults. Am J Addict. 2006;15 Suppl 1(Suppl 1):80-91. doi: 10.1080/10550490601006055. PMID 17182423
- [Background] Birchwood M, Smith J, Cochrane R, Wetton S, Copestake S. The Social Functioning Scale. The development and validation of a new scale of social adjustment for use in family intervention programmes with schizophrenic patients. Br J Psychiatry. 1990 Dec;157:853-9. doi: 10.1192/bjp.157.6.853. PMID 2289094
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addictions teachings hospital. — http://www.camh.ca/en/research/Pages/research.aspx

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Started | 23 | 41 | 46
4 Week Follow-Up | 16 | 33 | 33
Completed | 16 | 31 | 27
Not Completed | 7 | 10 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual | Total
Number analyzed (Participants) | 22 | 41 | 44 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.09 (15.79) | 36.44 (15.08) | 34.14 (14.20) | 34.60 (14.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 19 | 16 | 41
  Male | 16 | 22 | 28 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 17 | 39 | 41 | 97
  Unknown or Not Reported | 4 | 0 | 2 | 6
Education [Count of Participants; unit: Participants]
  High school not completed | 3 | 13 | 7 | 23
  High school completed | 6 | 12 | 11 | 29
  Post-secondary completed | 4 | 9 | 8 | 21
  Post-secondary attended | 8 | 6 | 18 | 32
  Unknown | 1 | 1 | 0 | 2
Not in a Relationship [Count of Participants; unit: Participants] | 18 | 35 | 37 | 90
Employment [Count of Participants; unit: Participants]
  Employed | 1 | 3 | 5 | 9
  Unemployed | 13 | 27 | 28 | 68
  Other Work Status | 8 | 11 | 10 | 29
  Unknown | 0 | 0 | 1 | 1
Number of Hospitalizations in the past year [Mean (Standard Deviation); unit: Hospitalizations] | 1.91 (1.48) | 1.54 (1.00) | 1.91 (1.43) | 1.76 (1.29)
Number of arrests in the past year [Number; unit: Arrests] | 1 | 5 | 5 | 11
Sexuality [Count of Participants; unit: Participants]
  Bisexual | 1 | 3 | 5 | 9
  Straight/Heterosexual | 18 | 34 | 33 | 85
  Other | 3 | 4 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Multnomah Community Ability Scale - Participant Interview Based
Description: Community Functioning and change in adaptive functioning will be assessed with the Multnomah Community Ability Scale (MCAS), a 17-item scale assessing domains of functionality including health, adjustment to living, social competence, and behavioral problems (completed at all time points). This measure best reflects the primary aim of this intervention: to support a greater degree of illness self-management, independence, and level of community activity. The MCAS will be scored based upon interviews with participants and by the primary clinician (inpatient for baseline and case managers for post and follow up measures). The total score is reported here and is the sum of the 4 subscale totals (Health, Adaptation, Social Skills, Behaviour). The min total score is 17 and the max is 85 with higher values representing better outcomes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 22 | 41 | 44
Total Score | 65.45 (15.67) | 67.83 (7.67) | 64.66 (11.81)

2. Primary Outcome: Multnomah Community Ability Scale - Participant Interview Based
Description: as for outcome 1
Time Frame: 4 Week Follow-Up
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 33 | 33
Total Score | 70.67 (2.08) | 71.04 (1.70) | 71.49 (1.20)

3. Primary Outcome: Multnomah Community Ability Scale - Participant Interview Based
Description: as for outcome 1
Time Frame: 6 Month Follow-Up
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 31 | 27
Total Score | 72.03 (2.43) | 68.65 (2.09) | 70.41 (1.6)

4. Primary Outcome: Multnomah Community Ability Scale - Clinician Based
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 22 | 41 | 44
Total Score | 63.05 (8.76) | 60.20 (14.14) | 60.11 (15.73)

5. Primary Outcome: Multnomah Community Ability Scale - Clinician Based
Description: as for outcome 1
Time Frame: 4 Week Follow-Up
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 33 | 33
Total Score | 60.15 (3.54) | 64.53 (2.89) | 65.99 (1.9)

6. Primary Outcome: Multnomah Community Ability Scale - Clinician Based
Description: as for outcome 1
Time Frame: 6 Month Follow-Up
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 31 | 27
Total Score | 66.64 (3.65) | 59.84 (3.07) | 65.97 (2.4)

7. Secondary Outcome: Hospitalizations and Emergency Room Visits
Description: The percentage of participants that were re-hospitalized or visited the emergency room during the study were captured through case manager report and verified through hospital electronic database if a CAMH hospitalization.
Time Frame: Baseline to 6 Month Follow-Up
Measure: Number; unit: percentage of participants in arm
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 22 | 41 | 44
percentage of participants in arm
  Hospitalizations | 13.6 | 12.2 | 6.8
  Emergency Room Visits | 13.6 | 7.3 | 9.1

8. Secondary Outcome: The Satisfaction With Life Scale
Description: Quality of Life will be assessed with the Satisfaction With Life scale, an 18-item scale comprised of 4 subscales assessing living situation (4 items), social relationships (6 items), work (2 items), self and present life (6 items). Items are rated from 0 (not at all) to 1 (very little) to 2 (average or OK) to 3 (a lot) to 4 (a great deal). Subscale scores are reported here. The min value for all subscales is 0. The max value for the Living Situation subscale is 16. The max value for both the Social Relationships subscale and the Self and Present Life subscale is 24. The max value for the Work subscale is 8. Higher subscale scores indicate better outcomes (i.e., greater satisfaction with that area of life).
Time Frame: 4 Week Follow-Up
Measure: Mean (Standard Error); unit: Subscale score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 33 | 33
Subscale score
  Living Situation Subscale | 2.31 (0.30) | 2.63 (0.24) | 2.70 (0.02)
  Social Relationships Subscale | 2.19 (0.28) | 2.14 (0.22) | 2.14 (0.15)
  Work Subscale | 1.94 (0.37) | 1.78 (0.30) | 1.74 (0.14)
  Self and Present Life Subscale | 2.44 (0.27) | 2.18 (0.22) | 2.36 (0.07)

9. Secondary Outcome: The Satisfaction With Life Scale
Description: as for outcome 8
Time Frame: 6 Month Follow-Up
Measure: Mean (Standard Error); unit: Subscale score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 31 | 27
Subscale score
  Living Situation Subscale | 2.66 (0.35) | 2.67 (0.29) | 2.23 (0.08)
  Social Relationships Subscale | 2.29 (0.33) | 2.22 (0.27) | 1.97 (0.04)
  Work Subscale | 1.87 (0.34) | 1.71 (0.28) | 1.63 (0.15)
  Self and Present Life Subscale | 2.45 (0.31) | 2.22 (0.26) | 2.28 (0.05)

10. Secondary Outcome: Social Support Survey
Description: Quality of Life will also be assessed using the Social Support Survey, a 19 item scale that measures emotional/information support, tangible support, affectionate support and positive social interaction. Overall support index (i.e., Total Score) is reported here and is calculated from averaging all items and then applying a transformation [i.e., minimum possible score subtracted from observed score (first difference) and maximum possible score (second difference) and then the first difference divided by the second difference and that quotient multiplied by 100] such that the min score is 0 and the max is 100. Higher scores indicate better outcomes (i.e., more frequent availability of different types of support).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 22 | 41 | 44
Total Score | 65.59 (20.69) | 64.07 (21.85) | 57.44 (18.58)

11. Secondary Outcome: Social Support Survey
Description: as for outcome 10
Time Frame: 4 Week Follow-Up
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 33 | 33
Total Score | 67.68 (4.99) | 60.54 (4.23) | 64.11 (2.9)

12. Secondary Outcome: Social Support Survey
Description: as for outcome 10
Time Frame: 6 Month Follow-Up
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 31 | 27
Total Score | 68.66 (6.24) | 63.54 (5.41) | 67.50 (3.9)

13. Secondary Outcome: Brief Symptom Inventory
Description: Changes in symptomatology will be assessed with the 53 item Brief Symptom Inventory (BSI); this widely used instrument has extensively demonstrated validity and reliability properties and assesses a wide range of symptom areas. Participants rank how distressing symptoms are from 0 (not at all) to 4 (a great deal). The 52 items are organized into 9 symptom dimensions: Somatization, Obsession-Compulsions, Interpersonal Sensitivity Items, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, and Psychoticism. Dimension scores are calculated by summing the values for the items included in that dimension and dividing by the number of items endorsed in that dimension. The Global Severity Index (GSI) is reported here. The GSI is calculated by summing all the dimensions plus four additional items and dividing by the total number of items responded to. The min value is 0 and the max value is 72. Higher scores indicate worse outcomes (i.e., more distressing symptoms).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Global Severity Index
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 22 | 41 | 44
Global Severity Index | 67.05 (49.39) | 62.41 (42.56) | 56.93 (38.19)

14. Secondary Outcome: Brief Symptom Inventory
Description: as for outcome 13
Time Frame: 4 Week Follow-Up
Measure: Mean (Standard Error); unit: Global Severity Index
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 33 | 33
Global Severity Index | 0.94 (0.16) | 0.77 (0.12) | 0.88 (0.11)

15. Secondary Outcome: Brief Symptom Inventory
Description: as for outcome 13
Time Frame: 6 Month Follow-Up
Measure: Mean (Standard Error); unit: Global Severity Index
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 31 | 27
Global Severity Index | 0.83 (0.22) | 0.93 (0.18) | 1.03 (0.17)

16. Secondary Outcome: Global Appraisal of Individual Needs (GAIN) - Short Screener Substance Disorder Subscale
Description: The 5-item Global Appraisal of Individual Needs Short Screener (GAIN-SS) Substance Disorder Subscale (5-items) will be used to measure common psychological, behavioral, and personal problems related to alcohol and drug use. Each item is rated from 4 to 0 with 4, 3 and 2 representing use or problems in the past month, 2-3 months ago and 4-12 months ago, respectively. Items rated 1 represent problems over a year ago and items rated 0 indicate never having that problem. The subscale score is the total number of responses that indicate substance use problems within the last year. Substance Disorder Subscale scores for each arm are reported here. The min value is 0 and the max value is 5. Higher scores indicate worse outcomes (i.e., more severe problems related to substance use).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Subscale score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 22 | 41 | 44
Subscale score | 1.23 (1.77) | 1.05 (1.47) | 1.88 (2.01)

17. Secondary Outcome: Global Appraisal of Individual Needs (GAIN) - Short Screener Substance Disorder Subscale
Description: as for outcome 16
Time Frame: 4 Week Follow-Up
Measure: Mean (Standard Error); unit: Subscale score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 33 | 33
Subscale score | 1.20 (0.37) | 1.25 (0.31) | 1.35 (0.99)

18. Secondary Outcome: Global Appraisal of Individual Needs (GAIN) - Short Screener Substance Disorder Subscale
Description: as for outcome 16
Time Frame: 6 Month Follow-Up
Measure: Mean (Standard Error); unit: Subscale score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 31 | 27
Subscale score | 1.24 (0.44) | 1.31 (0.37) | 1.51 (1.3)

19. Secondary Outcome: Personal Recovery Outcome Measure
Description: The brief, 10-item version of the Personal Recovery Outcome Measure was used to assess change in recovery engagement. Total score is reported here. Total score is calculated by summing all the responses. Min total score value is 0 and max total score value is 40. Higher scores indicate better outcomes (i.e., more engagement in recovery).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 22 | 41 | 44
Total Score | 26.64 (8.44) | 24.20 (7.97) | 25.23 (8.63)

20. Secondary Outcome: Personal Recovery Outcome Measure
Description: as for outcome 19
Time Frame: 4 Week Follow-Up
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 33 | 33
Total Score | 6.09 (0.44) | 6.48 (0.37) | 6.29 (1.5)

21. Secondary Outcome: Personal Recovery Outcome Measure
Description: as for outcome 19
Time Frame: 6 Month Follow-Up
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 31 | 27
Total Score | 6.61 (0.49) | 6.11 (0.42) | 6.22 (1.5)

22. Secondary Outcome: Community Integration Scale
Description: Community involvement will be assessed with the 11 item Community Integration Scale which was developed for the At Home study with a comparable population to assesses psychological and behavioural community engagement. The first 7 items measure physical integration (community presence) and the remaining 4 items measure psychological integration (sense of belonging). Community Involvement was assessed post intervention and at follow up and not during inpatient stay since it would not be valid due to contextual confounds with items. Total scores (i.e, the average of the responses) are reported here. The min total score value is -1 and the max is 2.5. Higher scores indicate better outcomes (i.e., greater community engagement)
Time Frame: 4 Week Follow-Up
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 33 | 33
Total Score | 1.44 (0.12) | 1.45 (0.10) | 1.31 (0.75)

23. Secondary Outcome: Community Integration Scale
Description: as for outcome 22
Time Frame: 6 Month Follow-Up
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
Number analyzed (Participants) | 16 | 31 | 27
Total Score | 1.39 (0.16) | 1.32 (0.13) | 1.49 (0.99)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Under "All Cause Mortality", the research team was notified of one participant death after the 6 month follow up assessment but prior to receiving the clinician-reported MCAS. As such, we counted them as still enrolled in the study at the time we were notified of their death.
Arm/Group | Welcome Basket Brief (WBbr) | Welcome Basket (WB) | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 0/22 | 2/41 | 0/44
Serious Adverse Events (participants affected / at risk) | 10/22 | 13/41 | 11/44
Other Adverse Events (participants affected / at risk) | 0/22 | 0/41 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Welcome Basket Brief (WBbr) (N=22) | Welcome Basket (WB) (N=41) | Treatment As Usual (N=44)
Hospitalizations (Inpatient) (Psychiatric disorders) | 10 | 13 | 11

LIMITATIONS AND CAVEATS:
The metrics employed in this study may have lacked sufficient sensitivity given the short time frame of this study. Other limitations of this study included its deployment at a single clinical site, a limited sample size, a relatively short follow-up period, and un-blinded participants. Diversity in participant clinical profiles and life circumstances may have also influenced these findings with a recruitment strategy that included both early intervention and chronic care units.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT02946255/Prot_SAP_000.pdf